CLINICAL TRIAL: NCT00763763
Title: Study to Evaluate Efficacy and Safety of Glivec® in Combination With Vincristine and Dexamethasone in Patients With Lymphoid Blast Crisis CML or Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia in Relapse or Refractory
Brief Title: Imatinib Mesylate With Vincristine and Dexamethasone in Acute Lymphoblastic Leukemias With BCR-ABL Positive
Acronym: AFR07
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P030425
Record Dates: First submitted 2008-07-25; First posted 2008-10-01 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Leukemia, Lymphocytic, Acute; Philadelphia Chromosome; Blast Crisis; Leukemia, Myeloid, Chronic
Keywords: Imatinib mesylate; Combination therapy; Leukemia, Lymphocytic, Acute; Philadelphia Chromosome; Blast Crisis; Leukemia, Myeloid, Chronic
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Philadelphia Chromosome; Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; Interferons; peginterferon alfa-2a; Vincristine; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): imatinib in combination with chemotherapy by vincristin and dexamethasone
  Interventions: Drug: Imatinib mesylate; Drug: Interferon; Drug: Vincristine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Imatinib mesylate — imatinib 600 mg/day for 2 years
  Other Names: Interferon, Pegasys
Drug: Interferon — 45 micrograms per week during 2 years
  Other Names: Pegasys
Drug: Vincristine — 2 mg IV injection repeated weekly for 4 weeks as induction and then monthly for 4 months as consolidation
Drug: Dexamethasone — 40 mg PO repeated weekly for 4 weeks as induction and then monthly for 4 months as consolidation

SUMMARY:
Patients not previously exposed to imatinib and with resistant or refractory Ph+ ALL, lymphoid blast crisis chronic myelogenous leukaemia (LBC CML) or with de novo Ph+ ALL and aged over 55y were eligible in the study. The DIV regimen consisted in one IV injection of vincristine 2 mg combined with 2 days of dexamethasone 40 mg PO repeated weekly for 4 weeks as induction and then monthly for 4 months as consolidation. Imatinib was administered at 800 mg per day during the induction period and at 600 mg/d continuously during consolidation. Patients in CR not eligible for HSCT were allocated to maintenance therapy consisting in weekly SC injection of Pegasys 45 µg and continuous administration of imatinib 400 mg per day for 2 years.

DETAILED DESCRIPTION:
Gleevec™ is now considered as the gold standard treatment in chronic phase chronic myeloid leukemia (CML), for patients who are not candidate for an allogenic bone marrow transplantation. However, in advanced phase CML and Philadelphia chromosome-positive acute lymphoblastic leukemia (Ph+ ALL), development of resistance to imatinib has become the central issue concerning the use of imatinib as a monotherapeutic agent. The response rate (complete hematological remission) at the dose of 600 mg/d in poor prognosis lymphoid blast phase CML and Ph+ ALL was about 20% and median time to disease progression was only 2.2 months. In VITRO studies have addressed the question of combined therapy with imatinib. A synergistic or additive activity has been demonstrated with vincristine and dexamethasone, two major drugs for the treatment of acute lymphoblastic leukemia (ALL). On going clinical studies are also testing Gleevec™ in association with daunorubicin and cytarabine (standard dose) in CML in myeloid blast phase (CST571AFR01) or with MITHOXANTROME and cytarabine (intermediate dose) as a consolidation regiment in Ph+ ALL in first CR (CSTI571AFR03). The safety of the combined therapy was excellent in the two studies. Therefore, we propose to initiate a study to assess the efficacy and the safety of Gleevec™ combined with vincristine and dexamethasone in patients with relapsed or refractory Philadelphia chromosome-positive acute lymphoblastic leukemias

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects over 18 years,
* Poor prognosis BCR-ABL transcript-positive acute lymphoblastic leukemia (refractory or relapsing Ph+ ALL, BP lymphoid CML, BP lymphoid CML in relapse)

Exclusion Criteria:

* Pregnant female,
* Blastic involvement of the CNS,
* Participation in an investigational agent trial within 4 weeks,
* High dose therapy within 4 weeks,
* Gleevec administration within 3 months,
* Transaminases grade 3 or 4 elevation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2004-12; Primary Completion 2007-10 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To determine the rate of hematological response induced by Gleevec™ combined with vincristine and dexamethasone | After 35 days or 56 days of induction

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ROUSSELOT, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Service Clinique des Maladies du Sang, Paris, Paris, France